CLINICAL TRIAL: NCT07285096
Title: Efficacy and Safety of P-CABs-Based Bismuth Quadruple Therapy for First-line Helicobacter Pylori Eradication: A Multicenter Cohort Study
Brief Title: P-CABs-based Bismuth Quadruple Therapy for Helicobacter Pylori Eradication
Acronym: PRO-HP
Status: Recruiting | Type: Observational
Sponsor: Yueyue Li (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Feicheng People's Hospital (Unknown); Binzhou Maternal and Child Health Hospital (Unknown); Jinxiang County People's Hospital (Unknown); The People's Hospital of Jimo (Unknown); Zibo Maternal and Child Health Hospital (Unknown); Yantai Penglai Traditional Chinese Medicine Hospital (Unknown); Zaozhuang Municipal Hospital (Other); Linyi Yizhou Hospital (Unknown); Taierzhuang District People's Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Yuncheng Traditional Chinese Medicine Hospital (Other); Caoxian County Hospital (Unknown); Qihe County People's Hospital (Unknown); University Town Hospital, Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Unknown); Dezhou Hospital Qilu Hospital of Shandong University (Other); The 2nd People's Hospital of Dongying City (Unknown); Zhangdian District Hospital of Traditional Chinese Medicine (Unknown); Yantai Zhifu Hospital (Unknown); Inner Mongolia Autonomous Region International Mongolian Medicine Hospital (Unknown); Hohhot Second Hospital (Unknown); Guanxian People's Hospital (Unknown); Longkou People's Hospital (Unknown); Linshu County Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Yueyue Li, Associate Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: 202511
Record Dates: First submitted 2025-11-27; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; quadruple therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vonoprazan-based quadruple therapies
  Interventions: Other: Doctors prescribe Helicobacter pylori treatment regimens for patients based on current guidelines and consensus statements, tailored to individual circumstances，not involve any intervention procedures
- tegoprazan-based quadruple therapies
  Interventions: Other: Doctors prescribe Helicobacter pylori treatment regimens for patients based on current guidelines and consensus statements, tailored to individual circumstances，not involve any intervention procedures

INTERVENTIONS:
Other: Doctors prescribe Helicobacter pylori treatment regimens for patients based on current guidelines and consensus statements, tailored to individual circumstances，not involve any intervention procedures — Doctors prescribe Helicobacter pylori treatment regimens for patients based on current guidelines and consensus statements, tailored to individual circumstances，not involve any intervention procedures.

SUMMARY:
Bismuth-containing quadruple therapy was recommended as a first-line treatment for Helicobacter pylori infection. This study aimed to compare real-world outcomes of various potassium-competitive acid blockers (P-CABs) -based bismuth quadruple regimens and identify factors influencing treatment failure. A multicenter cohort study was conducted and study outcomes included eradication rates and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-70 years, regardless of gender;
* willing to receive H. pylori eradication therapy;
* diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.

Exclusion Criteria:

* patients with incomplete medical records, including missing treatment details, absence of post-treatment follow-up test results, or failure to complete essential follow-up assessments;
* patients who received treatment regimens that did not comply with the quadruple regimens specified in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) patients aged 18-70 years, regardless of gender; (2) willing to receive H. pylori eradication therapy; (3) diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 1730 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 6-8 weeks after treatment completion
  Comparison of eradication rates among quadruple therapies for Helicobacter pylori

SECONDARY OUTCOMES:
Adverse events | lmmediately after treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China